CLINICAL TRIAL: NCT00419835
Title: Effect of Enalapril and Losartan Association Therapy on Proteinuria and Inflammatory Biomarkers in Diabetic Nephropathy: a Clinical Trial on Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST01
Record Dates: First submitted 2007-01-08; First posted 2007-01-09 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2007-01

CONDITIONS: Macroalbuminuric Diabetic Nephropathy
Keywords: diabetic nephropathy; proteinuria; CKD progression; dialysis
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria | interventions — Enalapril; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: enalapril
Drug: losartan

SUMMARY:
Chronic kidney disease (CKD)has become a significant health problem worldwide. Strategies to decrease the rate of progression of this disease and reduce the number of patients needing dialysis or renal transplantation are urgently needed. In this study we wish to compare the effect of dual blockade of renin-angiotensin system (ACE inhibitors plus angiotensin II receptor blocker) compared to the effect of ACE inhibitor monotherapy in patients with diabetic chronic nephropathy.

DETAILED DESCRIPTION:
Diabetic kidney disease is the current leading cause of chronic kidney disease (CKD) in the world. Despite all efforts to control this disease, rates of CKD progression are still high and a significant number of patients will ultimately need renal replacement therapy. Pharmacological blockade of renin-angiotensin system is one of the key elements of CKD secondary prevention, and ACE inhibitors or angiotensin II receptor 1 blocker (ARB)can be used for this purpose. However, it is still not clear if dual blockade (ACEi and ARBs simultaneously)is superior to monotherapy with ACE inhibitors or ARBs. A recent trial has suggested that dual blockade is superior to monotherapy in non-diabetic chronic kidney disease. The purpose of this trial is to evaluate the effect of combination therapy compared to ACE inhibitors alone in type 2 diabetic patients with macroalbuminuric diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* diabetic nephropathy characterised by a daily proteinuria superior to 500 mg
* type II diabetes

Exclusion Criteria:

* type 1 diabetes
* serum creatinine > 2.5 mg/dL or creatinine clearance lower than 30 ml/min
* serum potassium > 5.5 mEq/L
* intolerance or allergy to ACE inhibitors or BRA
* pregnancy
* hepatitis C or B
* HIV
* current chemotherapy treatment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
effect of treatment on proteinuria after 8 months of follow-up

SECONDARY OUTCOMES:
effect of treatment on urinary inflammatory biomarkers after 8 months of follow-up
incidence of hyperkalemia

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Zatz, Full Professor of Nephrology, Study Director — Nephrology Department, Sao Paulo University Medical School
Locations (1):
- Nephrology Department, Sao Paulo University Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Titan SM, Vieira JM Jr, Dominguez WV, Moreira SR, Pereira AB, Barros RT, Zatz R. Urinary MCP-1 and RBP: independent predictors of renal outcome in macroalbuminuric diabetic nephropathy. J Diabetes Complications. 2012 Nov-Dec;26(6):546-53. doi: 10.1016/j.jdiacomp.2012.06.006. Epub 2012 Sep 12. PMID 22981148
- [Derived] Titan SM, Zatz R, Graciolli FG, dos Reis LM, Barros RT, Jorgetti V, Moyses RM. FGF-23 as a predictor of renal outcome in diabetic nephropathy. Clin J Am Soc Nephrol. 2011 Feb;6(2):241-7. doi: 10.2215/CJN.04250510. Epub 2010 Oct 21. PMID 20966122